CLINICAL TRIAL: NCT04898829
Title: An Exploratory Study to Evaluate the Acceptability of PKU Explore, a Food for Special Medical Purposes, for Use in the Dietary Management of Phenylketonuria in Infants From 6 Months to 3 Years of Age With Regard to Product-acceptability, Tolerance, Phe Levels and Growth
Brief Title: Evaluation of PKU Explore France
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCT-W-PKUExp-2018-09-03; 2021-A00276-35 (Other: REC)
Record Dates: First submitted 2021-05-11; First posted 2021-05-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Phenylketonurias
Keywords: Phenylketonuria; PKU; Explore; France
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PKU Explore (Experimental): PKU Explore will be prescribed by the study dietitian based on the patient's individual requirement.
  Interventions: Dietary Supplement: PKU explore

INTERVENTIONS:
Dietary Supplement: PKU explore — For 28 consecutive days, participants will take their usual restricted therapeutic diet, either:
  - Replacing their usual second stage concentrated protein substitute with PKU explore
  OR
  - Commencing PKU explore and gradually reducing their Phe-free formula for infants.

SUMMARY:
PKU explore France is an exploratory study to evaluate the acceptability of PKU explore, a food for special medical purposes, for use in the dietary management of phenylketonuria in infants from 6 months to 3 years of age, assessing participant adherence, GI tolerance, phe levels, growth and product palatability.

DETAILED DESCRIPTION:
The study product, PKU explore, is a concentrated, spoonable, protein substitute food for special medical purposes, used in the dietary management of PKU. The recommended amount will be determined by a dietitian or clinician and the product used is unflavoured.

PKU explore France is an exploratory study to evaluate the gastrointestinal tolerance, palatability, and participant adherence over a four-week period in patients with PKU that follow an appropriate restricted therapeutic diet. This will be followed by a maximum 24-month follow-up period monitoring growth as per routine standard of care.

Up to 10 participants will be recruited at a single centre in France.

For 28 consecutive days, up to 10 participants, aged 6 months to 3 years inclusive, take their usual restricted therapeutic diet, either replacing their usual second-stage, concentrated protein substitute with PKU explore or commencing PKU explore and gradually reducing their Phe-free formula for infants.

Their parent/guardian complete a daily questionnaire on adherence and tolerance, and a final questionnaire on usage and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of PKU on new-born screening requiring a low protein diet and Phe-free L-amino acid protein substitute.
* Aged between 6 months and 3 years (inclusive at screening).
* Already taking part of their protein substitute in a spoonable form OR is at the stage in their PKU management when a second stage spoonable protein substitute is recommended to commence.
* Well-controlled PKU, evidenced by the latest three routine blood spots being within the acceptable range, in the investigator's opinion.
* Able to comply with the study protocol and take the study product, according to the opinion of the investigator.
* Willingly given, written, informed consent from parents/guardian.

Exclusion Criteria:

* Diagnosis of persistent hyperphenylalaninaemia, or mild PKU not requiring dietary intervention with a low protein diet and Phe-free L-amino acid supplements.
* Diagnosis of a concurrent condition which may adversely affect developmental progression and feeding ability.
* Known milk or fish allergy/intolerance.
* Patients who are currently participating in, plan to participate in or have participated in an interventional investigational drug, food or medical device trial within 30 days prior to the screening visit.
* Existing significant GI issues which may affect compliance with the study protocol, according to the opinion of the investigator.
* Any medical conditions precluding the study intervention, which in the opinion of the investigator may impact on metabolic control during the study period.
* Use of additional macro/micronutrient supplements during the study period, unless clinically indicated and prescribed by the investigator (must be recorded in patient case record file).
* Where applicable, patients NOT covered by Health Insurance System and/or not in compliance with the recommendations of National Law in force.

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Adherence to the recommended amount of study product | Days 1 - 28
  Quantitative assessments from subject questionnaires that allow evaluation of compliance with the study product (i.e. actual versus prescribed intake), measured in grams consumed per day.
Product palatability rated on a Likert scale by the patient after 28 days | Day 28
  Patient assessment of study product's palatability using a Likert scale. At the end of the 28-day acceptability phase, participants/parents/guardians will be required to complete a Product Acceptability Questionnaire to record perceptions about: the appearance, smell, taste, aftertaste, texture, packaging/presentation of the product, also the ease of preparation and administration.
  These will be on a 5-point Likert scale as Loved it, Liked it, Neither liked nor disliked it, Didn't like it and Really didn't like it.
Gastrointestinal tolerance daily diary as reported by the patient | Days 1 - 28
  Qualitative assessments from subject questionnaires to allow evaluation of any self-reported gastrointestinal symptoms during the study period.
Change in Phe levels | Previous three routine results prior to Visit 1, Visit 1 (Day 0), Week 1, Week 2, Week 3, Week 4 and Visit 2 (Day 28)
  Analysis of results from routine dried blood spots. Change in Phe level at diagnosis and at different timepoints measured as µmol/l.

SECONDARY OUTCOMES:
Evaluation of growth for a minimum of two years follow up period | Visit 1 (day 0), Visit 2 (Day 28) and Every 4 months for a max. 24 Months' Followup
  Height/length, weight and head circumference measurements will be combined to complete the growth chart at each visit. All recorded weights, lengths, and head circumferences will be plotted on a Croissance Somatique Des Garçons/Filles De La Naissance A 3 Ans Chart.
  The units of measurement are height/length in centimeters, weight in kilograms, and head circumference in centimeters.
Product adherence for a minimum of two years follow up period by measuring the quantity of product intake | days 1 - 28
  Measurement of the quantity of product intake. Quantitative assessments from subject questionnaires that allow evaluation of compliance with the study product, i.e. actual versus prescribed intake. Weight of powder prescribed per 24 hours in g (grams) and the number of feeds prescribed per 24 hours (feeds) will be recorded.
Product adherence for a minimum of two years follow up period by measuring the Phe levels | Visit 1 (Day 0), Week 1, Week 2, Week 3, Week 4, Visit 2 (Day 28) and every 4 months for a max. 24 Months' Follow-up period
  Measurement of phe levels in µmol/l throughout the evaluation period. The latest Phe level results will be recorded at each visit as µmol/l and compared.

CONTACTS AND LOCATIONS:
Overall Officials: Karine Mention, Principal Investigator — CHU Lille
Locations (1):
- Hôpital Jeanne de Flandre, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No